CLINICAL TRIAL: NCT04684524
Title: A Randomized Double-blind Placebo-controlled Parallel Group Study Assessing the Efficacy and Safety of Dupilumab in Patients With Allergic Fungal Rhinosinusitis (AFRS)
Brief Title: Dupilumab in Allergic Fungal Rhinosinusitis (AFRS) (LIBERTY-AFRS-AI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16724; U1111-1246-7549 (Registry Identifier: ICTRP); 2020-002999-12 (EudraCT Number)
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-11

CONDITIONS: Allergic Fungal Rhinosinusitis
MeSH Terms: conditions — Allergic Fungal Sinusitis | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): Dupilumab administered every 2 or 4 weeks based on weights
  Interventions: Drug: Dupilumab SAR231893
- Matching placebo (Placebo Comparator): Placebo administered every 2 or 4 weeks based on weights
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Dupilumab
Drug: Placebo — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Matching placebo

SUMMARY:
Primary Objective:

* To evaluate the efficacy of treatment with dupilumab to reduce sinus opacification in a population with allergic fungal rhinosinusitis (AFRS)

Secondary Objectives:

* To evaluate the efficacy of treatment with dupilumab to reduce sinus opacification in a population with allergic fungal rhinosinusitis (AFRS) at Week 24
* To assess the efficacy of dupilumab to reduce the need for rescue treatments
* To evaluate the efficacy of treatment with dupilumab in improving symptoms in AFRS
* To evaluate the efficacy of dupilumab to reduce nasal polyp formation in participants with AFRS
* To evaluate the efficacy of dupilumab in improving overall symptom severity and quality of life in AFRS
* To evaluate the efficacy of dupilumab in improving sense of smell in participants with AFRS
* To explore the effect of dupilumab as assessed by three-Dimensional CT volumetric measurement of the paranasal sinuses
* To evaluate the safety and tolerability of dupilumab when administered to participants with AFRS
* To evaluate the pharmacokinetics (PK) of dupilumab in participants with AFRS
* To characterize the effect of dupilumab on total IgE and specific IgE
* To assess immunogenicity to dupilumab in participants with AFRS

DETAILED DESCRIPTION:
The duration of study for each participant will include 2-4 weeks of screening period (2 additional weeks could be allowed), 52 weeks of randomized investigational medicinal product (IMP) intervention period and 12 weeks of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Participant must be at least 6 years of age (or the minimum legal age for adolescents in the country of the investigational site) at the time of signing the informed consent.

Participants with the diagnosis of AFRS adapted from criteria by Bent and Kuhn (meeting all):

* IgE mediated inflammatory response to fungal hyphae (specific IgE serology or skin test) Evidence of sensitization to fungus by skin testing (at screening or documented historical positive skin test in the previous 12 months), or positive fungal-specific IgE in serum at screening.
* Nasal polyposis confirmed by nasal endoscopy at screening.
* Characteristic CT signs to be performed during screening period and can include any of the below signs as assessed by central reader:

  * hyperdensities
  * bony demineralization
  * bone erosion of sinus
* Eosinophilic mucin/mucus identified within 5 years prior to screening or at screening with or without positive fungal stain

AFRS patients with the following:

* An endoscopic NPS of at least 2 out of 4 for unilateral polyps or 3 out of 8 for bilateral polyps at Visit 1 (central reading) and Visit 2 (local reading) and,
* Sinus opacification in CT scan with an LMK score of 9 for patients with unilateral polyps or 12 for patients with bilateral polyps during screening period and,

Body weight ≥15 kg

Exclusion Criteria:

* Patients with nasal conditions/concomitant nasal diseases making them non-evaluable at Visit 1 or for the primary efficacy
* Nasal cavity malignant tumor and benign tumors.
* Known of fungal invasion into sinus tissue.
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect the patient's participation in the study
* Active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis unless documented adequately treated.
* Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection
* Known or suspected immunodeficiency
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the Screening Visit 1 or during the screening period.
* History of systemic hypersensitivity or anaphylaxis to dupilumab or any of its excipients.
* Treatment with commercially available dupilumab within 12 months, participation in prior dupilumab clinical trial, or discontinued dupilumab use due to adverse event.
* Patients who are treated with intranasal corticosteroid drops; intranasal steroid emitting devices/stents; nasal spray using exhalation delivery system, such as Xhance™, during screening period.
* Patients who are on intranasal corticosteroids (INCS) spray unless they have received stable dose for at least 4 weeks prior to Visit 1.
* Patients who have undergone sinus intranasal surgery (including polypectomy) within 6 months prior to Visit 1.
* Patients who have taken:

  * Biologic therapy/systemic immunosuppressant to treat inflammatory disease or autoimmune disease within 5 half-lives prior to Visit 1
  * Any investigational mAb within 5 half-lives prior to Visit 1
  * Anti-IgE therapy (omalizumab) within 4 months prior to Visit 1. - Treatment with a live (attenuated) vaccine within 4 weeks prior to Visit 1
* Leukotriene antagonists/modifiers unless patient is on a continuous treatment for at least 30 days prior to Visit 1.
* Initiation of allergen immunotherapy within 3 months prior to Visit 1 or a plan to begin therapy or change its dose during the screening or treatment period. - Patients received SCS during screening period. - Either intravenous immunoglobulin therapy and/or plasmapheresis within 30 days prior to Screening Visit (Visit 1).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (47):
- United States (11):
  - Asthma Allergy & Immunology Clinical Research Unit Site Number : 8400001, Tampa, Florida
  - Emory University Hospital Midtown Campus Site Number : 8400009, Atlanta, Georgia
  - Advanced ENT and Allergy Site Number : 8400004, Louisville, Kentucky
  - South Louisiana Ear, Nose, Throat and Facial Plastic Surgery Site Number : 8400019, Mandeville, Louisiana
  - National Allergy and Asthma Research, LLC Site Number : 8400002, Charleston, South Carolina
  - Vanderbilt University Medical Center Site Number : 8400013, Nashville, Tennessee
  - REX Clinical Trials Site Number : 8400017, Beaumont, Texas
  - Ut- Houston Medical School Site Number : 8400010, Houston, Texas
  - USA Clinical Trials Site Number : 8400020, San Antonio, Texas
  - Alamo ENT Associates Site Number : 8400018, San Antonio, Texas
  - Eastern Virginia Medical School (EVMS) Medical Group - Otola Site Number : 8400008, Norfolk, Virginia
- Argentina (5):
  - Investigational Site Number : 0320003, CABA, Buenos Aires
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Mendoza
- Investigational Site Number : 1240001, Vancouver, British Columbia, Canada
- China (11):
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560004, Changsha
  - Investigational Site Number : 1560003, Chengdu
  - Investigational Site Number : 1560013, Fuzhou
  - Investigational Site Number : 1560006, Hangzhou
  - Investigational Site Number : 1560012, Hefei
  - Investigational Site Number : 1560002, Nanjing
  - Investigational Site Number : 1560011, Qingdao
  - Investigational Site Number : 1560009, Shanghai
  - Investigational Site Number : 1560008, Taiyuan
- India (3):
  - Investigational Site Number : 3560003, Coimbatore
  - Investigational Site Number : 3560006, Jodhpur
  - Investigational Site Number : 3560008, New Delhi
- Israel (2):
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760002, Rehovot
- Japan (6):
  - Investigational Site Number : 3920010, Isehara, Kanagawa
  - Investigational Site Number : 3920006, Shizuoka, Shizuoka
  - Investigational Site Number : 3920008, Bunkyo-ku, Tokyo
  - Investigational Site Number : 3920001, Meguro-ku, Tokyo
  - Investigational Site Number : 3920003, Shinagawa-ku, Tokyo
  - Investigational Site Number : 3920009, Shinjuku-ku, Tokyo
- Saudi Arabia (2):
  - Investigational Site Number : 6820002, Riyadh
  - Investigational Site Number : 6820001, Riyadh
- Turkey (Türkiye) (6):
  - Investigational Site Number : 7920004, Adana
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920007, Istanbul
  - Investigational Site Number : 7920006, Izmir
  - Investigational Site Number : 7920003, Izmir
  - Investigational Site Number : 7920005, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16724 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25253&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 45 centers in 9 countries. A total of 152 participants were screened from 01-Dec-2020 to 28-Nov-2023 of which 90 were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 62 participants were randomized in a 1:1 ratio to receive either dupilumab or matching placebo in this study. Reasons for study discontinuation are presented.
Groups:
- Placebo: Participants received placebo matched to dupilumab via subcutaneous (SC) injection for 52 weeks.
- Dupilumab: Participants received dupilumab depending on the weight at screening via SC injection for 52 weeks as follows:
  * 300 milligrams (mg) every 2 weeks (q2w) for all adults and adolescents/children weighing >=60 kilograms (kg)
  * 200 mg q2w for adolescents/children weighing >=30 kg and <60 kg
  * 300 mg every 4 weeks (q4w) for adolescents/children weighing >=15 kg and <30 kg.
Period: Overall Study
Arm/Group | Placebo | Dupilumab
Started | 29 | 33
Randomized and Treated | 28 | 33
Completed | 21 | 29
Not Completed | 8 | 4
Not completed — Other | 2 | 0
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which included all participants from screened population who were allocated to a randomized drug by interactive response technology regardless of whether the drug was received or not.
Groups:
- Placebo: Participants received placebo matched to dupilumab via SC injection for 52 weeks.
- Dupilumab: Participants received dupilumab depending on the weight at screening via SC injection for 52 weeks as follows:
  * 300 mg q2w for all adults and adolescents/children weighing >=60 kg
  * 200 mg q2w for adolescents/children weighing >=30 kg and <60 kg
  * 300 mg q4w for adolescents/children weighing >=15 kg and <30 kg.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab | Total
Number analyzed (Participants) | 29 | 33 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (14.0) | 41.9 (17.5) | 39.8 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 13 | 17
  Male | 25 | 20 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 5 | 8
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Lund Mackay (LMK) score [Mean (Standard Deviation); unit: score on a scale] — LMK total score is based on assessment of computerized tomography (CT) scan findings for each sinus area (maxillary, anterior ethmoid, posterior ethmoid, sphenoid and frontal sinus plus osteomeatal complex on each side).Extent of sinus opacification is rated on 3-point scale; range 0 = normal to 2 = total opacification.In addition, osteomeatal complex is graded as 0 = not occluded or 2 = occluded.Maximum score is 12 per side; total score ranges from 0(normal) to 24(more opacified) corresponding to sum of all sinuses and osteomeatal complexes bilaterally.Higher score indicated worse outcome.
  score on a scale | 18.4 (3.4) | 17.5 (3.8) | 17.9 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 52 in Opacification of Sinuses Assessed by CT Scan Using the LMK Score
Description: The LMK score is used to quantify the degree of opacification of each sinus on CT scan. The CT scan LMK staging system represents the most widely established method of sinus CT scoring. The LMK total score is based on assessment of the CT scan findings for each sinus area (maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal sinus plus the osteomeatal complex on each side). The extent of sinus opacification is rated on a 3-point scale ranging from 0 = normal to 2 = total opacification. In addition, the osteomeatal complex is graded as 0 = not occluded or 2 = occluded. The maximum score is 12 per side; total score ranges from 0 (normal) to 24 (more opacified) corresponding to the sum of all sinuses and the osteomeatal complexes bilaterally. Higher score indicate worse outcome; a negative change from baseline indicate improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 52
Population: The intent-to-treat (ITT) population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -1.81 (0.81) | -9.17 (0.74)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Each of the imputed complete data were analyzed by fitting an analysis of covariance (ANCOVA) model with the corresponding baseline value, intervention group, time from last surgery (<=2 years, >2 years), and region (Americas and Asia) as covariates; Test type: Superiority; p < 0.0001, ANCOVA; Least squares (LS) Mean Difference = -7.36, 95% CI 2-sided [-9.38 to -5.35]

2. Secondary Outcome: Change From Baseline to Week 24 in Monthly Average Nasal Congestion/Obstruction Score From the Nasal Symptom Diary
Description: The nasal symptom diary is designed to assess the severity of chronic rhinosinusitis (CRS) nasal symptoms on daily basis. Score range: 0 = no symptoms, 1 = mild symptoms (symptoms clearly present, but minimal awareness and easily tolerated), 2= moderate symptoms (definite awareness of symptoms that is bothersome but tolerable) and 3 = severe symptoms (symptoms that are hard to tolerate, cause interference with activities or daily living). Higher scores denote greater symptom severity; a negative change from baseline indicate improvement. Baseline was defined as the average of the scores in the 7 days prior to the first dose of study drug.
Time Frame: Baseline (Day -7 to Day -1) and Week 24
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.43 (0.13) | -1.30 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Each of the imputed complete data were analyzed by fitting an ANCOVA model with the corresponding baseline value, intervention group, time from last surgery (<=2 years, >2 years), and region (Americas and Asia) as covariates; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.87, 95% CI 2-sided [-1.18 to -0.56]

3. Secondary Outcome: Change From Baseline to Week 24 in Endoscopy Nasal Polyp Score (NPS)
Description: The bilateral endoscopy NPS is determined by the clinician who assesses nasal polyp formation. Polyps on each side of the nose are graded based on polyp size; scores: 0 = no polyps; 1 = small polyps in the middle meatus not reaching below the inferior border of the middle turbinate; 2 = polyps reaching below the lower border of the middle turbinate; 3 = large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate and 4 = large polyps causing complete obstruction. The total score is the sum of the right and left nostrils, ranging from 0 (no obstruction) to 8 (complete obstruction); higher score indicating worse outcome; a negative change from baseline indicate improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.80 (0.38) | -3.16 (0.34)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.36, 95% CI 2-sided [-3.31 to -1.41]

4. Secondary Outcome: Change From Baseline to Week 24 in Opacification of Sinuses Assessed by CT Scan Using the LMK Score
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -1.93 (0.82) | -7.38 (0.80)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -5.45, 95% CI 2-sided [-7.48 to -3.43]

5. Secondary Outcome: Change From Baseline to Week 24 in Monthly Average Total Symptom Score (TSS) Derived From the Nasal Symptom Diary
Description: The nasal symptom diary is designed to assess the severity of CRS nasal symptoms on daily basis. The TSS is a composite score consisting of the sum of the following symptoms assessed daily in the morning: nasal congestion/obstruction, decreased/loss of sense of smell, rhinorrhea (average of anterior/posterior nasal discharge). Each of the individual items were scored from 0 = no symptoms to 3 = severe symptoms. TSS is the sum of individual items and ranges between 0 = no symptoms and 9 = severe symptoms. Higher scores on the TSS indicate greater symptom severity; a negative change from baseline indicate improvement. Baseline was defined as the average of the scores in the 7 days prior to the first dose of study drug.
Time Frame: Baseline (Day -7 to Day -1) and Week 24
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -1.26 (0.35) | -3.45 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.18, 95% CI 2-sided [-3.04 to -1.32]

6. Secondary Outcome: Change From Baseline to Week 24 in University of Pennsylvania Smell Identification Test (UPSIT)
Description: The UPSIT (UPSIT 40 odorant test) is a rapid and easy-to-administer method to quantitatively assess human olfactory function. The test consists of 4 booklets, each containing 10 odorants with 1 odorant per page. Above each odorant strip is a multiple-choice question with 4 alternative words to describe the odor and the participant is asked to indicate which word best describes the odor. Each smell has a possible of 4 answers with one being correct, therefore the potential total scores can range from 0 (worst possible score) to 40 (best possible score), with 1 point being awarded for each correctly identified odor. Scores of <=18 were classified as anosmia, 19 to 25 as severe microsmia, 26 to 30 as moderate microsmia, 31 to 34 as mild microsmia, and 35 to 40 as normal smell appreciation. Higher scores indicated better olfactory function; i.e. better sense of smell. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | 4.41 (1.71) | 8.87 (1.60)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0392, ANCOVA; LS Mean Difference = 4.46, 95% CI 2-sided [0.22 to 8.71]

7. Secondary Outcome: Change From Baseline to Week 24 in Monthly Average Decreased/Loss of Smell Using the Nasal Symptom Diary
Description: The nasal symptom diary is designed to assess the severity of CRS nasal symptoms on daily basis. Decreased/loss of smell is scored as: 0 = no symptoms, 1 = mild symptoms (symptoms clearly present, but minimal awareness and easily tolerated), 2= moderate symptoms (definite awareness of symptoms that is bothersome but tolerable) and 3 = severe symptoms (symptoms that are hard to tolerate, cause interference with activities or daily living). Higher scores denote greater symptom severity; a negative change from baseline indicate improvement. Baseline was defined as the average of the scores in the 7 days prior to the first dose of study drug.
Time Frame: Baseline (Day -7 to Day -1) and Week 24
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.39 (0.16) | -1.28 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -0.89, 95% CI 2-sided [-1.29 to -0.49]

8. Secondary Outcome: Change From Baseline to Week 52 in Endoscopy NPS
Description: as for outcome 3
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.55 (0.43) | -3.32 (0.39)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.77, 95% CI 2-sided [-3.82 to -1.72]

9. Secondary Outcome: Change From Baseline to Week 52 in Monthly Average Nasal Congestion/Obstruction Score From the Nasal Symptom Diary
Description: The nasal symptom diary is designed to assess the severity of CRS nasal symptoms on daily basis. Score range: 0 = no symptoms, 1 = mild symptoms (symptoms clearly present, but minimal awareness and easily tolerated), 2= moderate symptoms (definite awareness of symptoms that is bothersome but tolerable) and 3 = severe symptoms (symptoms that are hard to tolerate, cause interference with activities or daily living). Higher scores denote greater symptom severity; a negative change from baseline indicate improvement. Baseline was defined as the average of the scores in the 7 days prior to the first dose of study drug.
Time Frame: Baseline (Day -7 to Day -1) and Week 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.17 (0.15) | -1.57 (0.14)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -1.40, 95% CI 2-sided [-1.77 to -1.02]

10. Secondary Outcome: Change From Baseline to Week 52 in 22-item Sino-Nasal Outcome Test (SNOT-22) Total Score
Description: The SNOT-22 is a validated questionnaire designed to assess the impact of CRS on participants health-related quality of life (HRQoL) and has 22 items covering symptoms, social/emotional impact, productivity, and sleep consequences of CRS. The recall period is past 2 weeks. Each item is rated on a 6-point Likert scale; response options ranging from 0 = no problem to 5 = problem as bad as it can be. A global score ranging from 0 (no impact) to 110 (severe impact) is calculated by summing the responses to all items; higher score indicates greater rhinosinusitis-related health burden; a negative change from baseline indicate improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all randomized participants. Only those participants with data collected at baseline and Week 52 are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 28 | 33
score on a scale | -12.64 (4.06) | -29.94 (3.75)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0004, ANCOVA; LS Mean Difference = -17.30, 95% CI 2-sided [-26.86 to -7.74]

11. Secondary Outcome: Change From Baseline to Week 52 in Three-dimensional CT Total Volume Occupied by Disease in All Sinuses
Description: This method is used to calculate the percent occupied by disease. It is performed at locations including ethmoid sinus, frontal sinus, maxillary sinus, and sphenoid sinus. The total volume occupied by disease in all sinuses is reported here. For the analysis, central reading at baseline was used for comparison with Week 52 reading. It is graded on a scale of 0-100%; a higher score is worse and indicates greater volume occupied by disease. A negative change from baseline indicated improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
percent | -5.73 (3.91) | -42.04 (3.47)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -36.31, 95% CI 2-sided [-45.59 to -27.03]

12. Secondary Outcome: Percentage of Participants Who Received Systemic Corticosteroids (SCS) and/or Underwent or Planned to Undergo Surgery for Allergic Fungal Rhinosinusitis (AFRS) at Week 52
Description: SCS use was defined as the use of SCS for rescue treatment of AFRS or for another reason and was captured by the Investigator (or designee) in electronic case report form (eCRF). Participants who underwent or planned to undergo surgery for AFRS were also recorded in eCRF.
Time Frame: Week 52
Population: The ITT population included all randomized participants.
Measure: Number; unit: percentage of particpants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
percentage of particpants | 31.0 | 3.0
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; Risk difference was estimated using Mantel-Haenszel estimate and confidence limits, with Mantel-Haenszel stratum weights for time from last surgery (<=2 years, >2 years) and region (Americas and Asia) and the Sato variance estimator; Test type: Superiority; p = 0.0010, Mantel Haenszel; Risk Difference (RD) = -29.1, 95% CI 2-sided [-46.42 to -11.79]

13. Secondary Outcome: Change From Baseline to Week 24 in SNOT-22 Total Score
Description: The SNOT-22 is a validated questionnaire designed to assess the impact of CRS on participants HRQoL and has 22 items covering symptoms, social/emotional impact, productivity, and sleep consequences of CRS. The recall period is past 2 weeks. Each item is rated on a 6-point Likert scale; response options ranging from 0 = no problem to 5 = problem as bad as it can be. A global score ranging from 0 (no impact) to 110 (severe impact) is calculated by summing the responses to all items; higher score indicates greater rhinosinusitis-related health burden; a negative change from baseline indicate improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 24
Population: The ITT population included all randomized participants. Only those participants with data collected at baseline and Week 24 are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 28 | 33
score on a scale | -11.63 (4.02) | -26.74 (3.81)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0032, ANCOVA; LS Mean Difference = -15.11, 95% CI 2-sided [-25.15 to -5.07]

14. Secondary Outcome: Percent Change From Baseline in Serum Total Immunoglobulin-E (IgE) to Week 52
Description: Blood samples were collected at specified timepoints for the assessment of IgE. Total IgE was measured with a quantitative method approved for diagnostic testing; a negative change from baseline indicate improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 52
Population: The safety population included all randomized participants who took at least 1 dose of study drug, regardless of the amount of treatment administered.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 28 | 33
percent change | 6.91 (10.86) | -73.81 (11.40)
Statistical Analysis 1: Comparison: Placebo vs Dupilumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -80.72, 95% CI 2-sided [-112.82 to -48.61]

15. Secondary Outcome: Change From Baseline to Weeks 24 and 52 in the Monthly Average Rhinorrhea Score From the Nasal Symptom Diary
Description: The nasal symptom diary is designed to assess the severity of CRS nasal symptoms on daily basis. Score range: 0 = no symptoms, 1 = mild symptoms (symptoms clearly present, but minimal awareness and easily tolerated), 2= moderate symptoms (definite awareness of symptoms that is bothersome but tolerable) and 3 = severe symptoms (symptoms that are hard to tolerate, cause interference with activities or daily living). Higher scores denote greater symptom severity; a negative change from baseline indicate improvement. Severity of rhinorrhea (average of anterior [runny nose]/posterior nasal discharge [post-nasal drip]) is presented here. Baseline was defined as the average of the scores in the 7 days prior to the first dose of study drug.
Time Frame: Baseline (Day -7 to Day -1) and Weeks 24 and 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale
  Week 24 | -0.44 (0.13) | -0.92 (0.12)
  Week 52 | -0.33 (0.15) | -1.09 (0.13)

16. Secondary Outcome: Change From Baseline to Week 52 in Monthly Average TSS Derived From the Nasal Symptom Diary
Description: as for outcome 5
Time Frame: Baseline (Day -7 to Day -1) and Week 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.71 (0.39) | -4.10 (0.35)

17. Secondary Outcome: Change From Baseline to Weeks 24 and 52 in Visual Analog Scale (VAS) Rhinosinusitis
Description: The rhinosinusitis VAS is used to evaluate the overall severity of the rhinosinusitis. It is a recommended scale to determine the participant's disease severity and to guide the treatment for CRS. The participant is asked to answer the following question: "How troublesome are your symptoms of your rhinosinusitis" on a 10-centimeter VAS from 0 = not troublesome to 10 = worst thinkable troublesome. Based on their score on the VAS, the severity of rhinosinusitis is divided into 3 categories as follows: mild = VAS 0 to 3, moderate = VAS >3 to 7 and severe = VAS >7 to 10; higher score indicating worse outcome; a negative change from baseline indicate improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Weeks 24 and 52
Population: The ITT population included all randomized participants. Only those participants with data collected at specified timepoints are reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 28 | 33
score on a scale
  Week 24 | -1.29 (0.61) | -4.30 (0.58)
  Week 52 | -1.20 (0.57) | -5.52 (0.54)

18. Secondary Outcome: Change From Baseline to Week 52 in UPSIT
Description: The UPSIT (UPSIT 40 odorant test) is a rapid and easy-to-administer method to quantitatively assess human olfactory function. The test consists of 4 booklets, each containing 10 odorants with 1 odorant per page. Above each odorant strip is a multiple-choice question with 4 alternative words to describe the odor and the participant is asked to indicate which word best describes the odor. Each smell has a possible of 4 answers with one being correct, therefore the potential total scores can range from 0 (worst possible score) to 40 (best possible score), with 1 point being awarded for each correctly identified odor. Scores of <=18 were classified as anosmia, 19 to 25 as severe microsmia, 26 to 30 as moderate microsmia, 31 to 34 as mild microsmia, and 35 to 40 as normal smell appreciation. Higher scores indicated better olfactory function, i.e. better sense of smell. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | 2.12 (1.73) | 9.45 (1.57)

19. Secondary Outcome: Change From Baseline to Week 52 in Monthly Average Decreased/Loss of Smell Using the Nasal Symptom Diary
Description: as for outcome 7
Time Frame: Baseline (Day -7 to Day -1) and Week 52
Population: The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 29 | 33
score on a scale | -0.24 (0.17) | -1.41 (0.16)

20. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or was a medically important event. TEAEs were AEs that developed, worsened or became serious during the treatment-emergent period.
Time Frame: From first dose of study drug (Day 1) up to end of follow-up per participant, up to approximately 64 weeks
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 28 | 33
Participants
  TEAEs | 22 | 23
  TESAEs | 3 | 0

21. Secondary Outcome: Serum Concentration of Dupilumab Over Time
Description: Blood samples were collected at the specified timepoints to obtain serum concentration of dupilumab.
Time Frame: Baseline (Day 1) and Weeks 12, 24 and 52
Population: The pharmacokinetic (PK) population included all participants in the safety population with at least 1 post-baseline PK result. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | Dupilumab
Number analyzed (Participants) | 19
nanogram/milliliter
  Day 1: number analyzed (Participants) | 13
  Day 1 | 0.00 (0.00)
  Week 12: number analyzed (Participants) | 14
  Week 12 | 47750.00 (17828.70)
  Week 24: number analyzed (Participants) | 18
  Week 24 | 49597.78 (26542.80)
  Week 52 | 57284.21 (27401.32)

22. Secondary Outcome: Percent Change From Baseline in Fungal-specific IgE at Week 52
Description: Blood samples were collected at specified timepoints for the assessment of fungal-specific IgE which was measured with a quantitative method approved for diagnostic testing; a negative change from baseline indicated improvement. Baseline was defined as the last available value before the first dose of study drug.
Time Frame: Baseline (Day 1) and Week 52
Population: The safety population included all randomized participants who took at least 1 dose of study intervention, regardless of the amount of treatment administered. Only those participants with data collected at Baseline and Week 52 are reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 15 | 13
percent change
  A. fumigatus Antigen IgE Antibody (AB): number analyzed (Participants) | 1 | 3
  A. fumigatus Antigen IgE Antibody (AB) | -65.79 | -77.20 (9.00)
  F. proliferatum Antigen IgE AB: number analyzed (Participants) | 11 | 10
  F. proliferatum Antigen IgE AB | -20.18 (38.03) | -66.09 (16.88)
  C. lunata Antigen IgE AB: number analyzed (Participants) | 12 | 10
  C. lunata Antigen IgE AB | 1.56 (29.80) | -74.82 (12.34)
  S. rostrata Antigen IgE AB: number analyzed (Participants) | 12 | 10
  S. rostrata Antigen IgE AB | 28.89 (52.58) | -61.77 (14.37)
  C. albicans Antigen IgE AB: number analyzed (Participants) | 14 | 13
  C. albicans Antigen IgE AB | 15.69 (33.17) | -63.60 (17.06)
  B. spicifera Antigen IgE AB: number analyzed (Participants) | 12 | 10
  B. spicifera Antigen IgE AB | 19.12 (52.10) | -56.26 (22.36)
  A. niger Antigen IgE AB: number analyzed (Participants) | 8 | 8
  A. niger Antigen IgE AB | 2.46 (55.43) | -67.48 (13.72)
  A. flavus Antigen IgE AB: number analyzed (Participants) | 11 | 9
  A. flavus Antigen IgE AB | 0.75 (44.77) | -52.94 (19.62)
  A. tenuis alternata Antigen IgE AB: number analyzed (Participants) | 15 | 11
  A. tenuis alternata Antigen IgE AB | 16.06 (47.96) | -56.07 (21.78)
  Mould Mix 2 IgE: number analyzed (Participants) | 5 | 8
  Mould Mix 2 IgE | -17.50 (29.93) | -66.81 (20.86)

23. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibodies (ADA) to Dupilumab
Description: Plasma samples were collected to evaluate antibodies to dupilumab. Treatment-emergent ADA responses were defined as a positive response in the ADA assay post first dose, when baseline results were negative or missing.
Time Frame: From first dose of study drug (Day 1) up to end of follow-up per participant, up to approximately 64 weeks
Population: The ADA population included all participants from the safety population with at least 1 post-baseline ADA result (positive, negative or inconclusive).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab
Number analyzed (Participants) | 19 | 22
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events and deaths were assessed from first dose of study drug (Day 1) up to end of follow-up per participant, up to approximately 64 weeks
Description: Analysis was performed on the safety population.
Arm/Group | Placebo | Dupilumab
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/28 | 0/33
Other Adverse Events (participants affected / at risk) | 15/28 | 16/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Dupilumab (N=33)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Allergic Fungal Rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Dupilumab (N=33)
Covid-19 (Infections and infestations) | 4 (4) | 5 (5)
Suspected Covid-19 (Infections and infestations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Allergic Fungal Rhinosinusitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04684524/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04684524/SAP_001.pdf